CLINICAL TRIAL: NCT01165346
Title: Stereotaxic Irradiation of Hepatocellular Carcinoma : Phase II Study
Brief Title: Stereotaxic Irradiation of Hepatocellular Carcinoma
Acronym: CKNO-HEP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CKNO-HEP-0703
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: liver cancer; hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Fiducial Markers; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotaxic radiation by CyberKnife (Experimental): Implantation of fiducials Stereotaxic radiation by CyberKnife : 3 X 15 Gy over 8 to 10 days
  Interventions: Radiation: Fiducials; Radiation: CyberKnife

INTERVENTIONS:
Radiation: Fiducials — Implantation of fiducials
Radiation: CyberKnife — 3 fractions over 8 to 10 days, 15 Gy/fraction

SUMMARY:
Stereotaxic radiation by CyberKnife : 3 X 15 Gy over 8 to 10 days for a total of 45 Gy.

DETAILED DESCRIPTION:
Stereotaxic radiation by CyberKnife : 3 X 15 Gy over 8 to 10 days for a total of 45 Gy

ELIGIBILITY:
Inclusion Criteria:

* Primitive liver cancer (hepatocellular carcinoma), proved by histology or diagnostic according to BCLC criteria
* T1-3 N0 M0
* With only one intra hepatic lesion and dimensions between 1 cm and 6 cm (IRM or hepatic scanner)
* Stereotaxic radiotherapy treatment approved in multidisciplinary consultation, the patient being rejected for standard therapeutic
* Age >= 18 ans
* Previous anti tumoral treatment allowed but suspended since at least 15 days before the inclusion
* OMS =< 2
* Portal thrombosis allowed
* Portal high blood pressure allowed
* No contraindication of fiducials implantation, hemostasis disorders must be treated before the implantation
* In case of underlying cirrhosis, only the Child-Pugh A is allowed
* Life expectancy >= 12 weeks
* Women must have an active contraception during all the study
* Patient affiliated to health insurance
* Patient must sign the consent

Exclusion Criteria:

* T4
* Cirrhosis Child B and C
* Hepatic lesion < 1 cm or > 6 cm
* 2 hepatic lesions or more
* Recurrent or metastatic disease
* Patient already included in another therapeutic trial with an experimental molecule
* Allergy to gold
* Pregnant women or susceptible to be pregnant or breastfeeding
* Unable for medical follow-up (geographic, social or mental reasons)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-08-31 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2018-04-19 (Actual)

PRIMARY OUTCOMES:
non-progression part | Up to 18 months
  Percentage of non-progression 18 months after treatment, according to RECIST criteria

SECONDARY OUTCOMES:
acute and late tolerance | Up to 5 years after treatment
  Evaluation of acute tolerance during 90 days after treatment and late tolerance after 90 days, according to NCI CTCAE v3.0 and RTOG criteria.
hepatic non progression part | Up to 3, 6, 9, 12 months
  Percentage of hepatic non progression at 3, 6, 9, 12 months of treatment, according to RECIST criteria.
median time without progression | Up to 5 years after treatment
  Time between :
  * Date of inclusion
  * Date of progression
Best response | Up to 5 years after treatment
  determination of the best response of treatment, according to RECIST
tumor evaluation | Up to 5 years after treatment
  According to EASL
Quality of life | Up to 18 months after treatment
  Questionnaire EORTC QLQ-C30 and QLQ-HCC18
Biological response | Up to 3, 6, 9 months
  tumoral marker : Alpha-fetoprotein
Medical costs | During the first 3 months
  micro-costing

CONTACTS AND LOCATIONS:
Overall Officials: Xavier MIRABEL, MD, Principal Investigator — Centre Oscar Lambret
Locations (4):
- France (4):
  - Centre François Baclesse, Caen
  - Centre Oscar LAMBRET, Lille
  - Centre Léon Bérard, Lyon
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No